CLINICAL TRIAL: NCT01793259
Title: An Open-label, Randomized, Two-period Cross-over Study of Repeated Subcutaneous Injections of Methotrexate 50mg/ml Solution Either by a Pre-filled Syringe (Reference) or by a Disposable Pre-filled Pen (Test) to Assess Patient's Preference and Self-injection Experience and to Compare the Local Tolerability in Patients With Active Rheumatoid Arthritis
Brief Title: Preference Methotrexate (MTX) Pre-filled Syringe Versus Pre-filled Pen in Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: medac GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MC-MTX.11/RA
Record Dates: First submitted 2013-02-14; First posted 2013-02-15 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- prefilled pen then prefilled syringe (Other): weekly methotrexate injection with a prefilled pen during 3 weeks and subsequently with the prefilled syringe the last 3 weeks
  Interventions: Drug: methotrexate prefilled pen; Drug: methotrexate prefilled syringe
- prefilled syringe then prefilled pen (Other): weekly methotrexate injection with a prefilled syringe during 3 weeks and subsequently with the prefilled pen the last 3 weeks
  Interventions: Drug: methotrexate prefilled pen; Drug: methotrexate prefilled syringe

INTERVENTIONS:
Drug: methotrexate prefilled pen
Drug: methotrexate prefilled syringe

SUMMARY:
The primary objective of this study is to assess the number of patients preferring the methotrexate pre-filled pen to the methotrexate pre-filled syringe after 6 weeks of treatment based on a questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age between 18 and 75 years
* Rheumatoid arthritis according to the American College of Rheumatology (ACR) criteria 1987 or ACR/European Liga Against Rheumatology (EULAR)2010
* Disease activity score (DAS) 28 > 2.6

Main Exclusion Criteria:

* Prior or other current subcutaneous treatment with self-injection
* Prior or concomitant treatment with biologics
* Contraindications to MTX treatment
* History or diagnosis of a dermatological disease at the injection site
* Women with child-bearing potential who do not use a highly effective method of contraception or men who have a partner with child-bearing potential and do not use a contraception during the study and at least 6 months thereafter.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-07; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
number of patients preferring the MTX pre-filled pen to the pre-filled syringe | after 6 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Müller-Ladner, MD, Principal Investigator — Kerckoff clinic, Bad Nauheim, Germany
Locations (1):
- Kerckhoff Clinic, Bad Nauheim, Germany

REFERENCES:
- [Derived] Demary W, Schwenke H, Rockwitz K, Kastner P, Liebhaber A, Schoo U, Hubner G, Pichlmeier U, Guimbal-Schmolck C, Muller-Ladner U. Subcutaneously administered methotrexate for rheumatoid arthritis, by prefilled syringes versus prefilled pens: patient preference and comparison of the self-injection experience. Patient Prefer Adherence. 2014 Aug 6;8:1061-71. doi: 10.2147/PPA.S64111. eCollection 2014. PMID 25125973